CLINICAL TRIAL: NCT07195734
Title: A Phase II Randomized Trial of Neoadjuvant Chemotherapy or Chemo-Immunotherapy in Patients With Recurrent/Persistent PD-L1 Enriched Squamous Cell Carcinoma of the Head and Neck Undergoing Salvage Surgery (NEOPOLIS)
Brief Title: Testing the Addition of Chemotherapy or Chemo-Immunotherapy to the Usual Surgery for Advanced Head and Neck Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-06920; NCI-2025-06920 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-HN015 (Other: NRG Oncology); NRG-HN015 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2025-09-26; First posted 2025-09-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Clinical Stage II HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Locally Recurrent Head and Neck Squamous Cell Carcinoma; Locally Recurrent Hypopharyngeal Squamous Cell Carcinoma; Locally Recurrent Laryngeal Squamous Cell Carcinoma; Locally Recurrent Oral Cavity Squamous Cell Carcinoma; Locally Recurrent Oropharyngeal Squamous Cell Carcinoma; Stage II Laryngeal Cancer AJCC v8; Stage II Lip and Oral Cavity Cancer AJCC v8; Stage II Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage III Laryngeal Cancer AJCC v8; Stage III Lip and Oral Cavity Cancer AJCC v8; Stage III Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVA Laryngeal Cancer AJCC v8; Stage IVA Lip and Oral Cavity Cancer AJCC v8; Stage IVA Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVB Laryngeal Cancer AJCC v8; Stage IVB Oropharyngeal (p16-Negative) Carcinoma AJCC v8
MeSH Terms: conditions — Oropharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Carcinoma | interventions — Specimen Handling; Carboplatin; cemiplimab; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Paclitaxel; Taxes; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (Salvage surgery) (Active Comparator): Patients undergo standard of care salvage surgery. Starting within 8 weeks of surgery, patients with high risk features also undergo radiation therapy daily for 5 treatments per week for 6 weeks and receive cisplatin IV once per week for 6 weeks during radiation treatment, in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, PET scan and optionally undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Procedure: Salvage Surgery
- Arm 2 (Chemotherapy, salvage surgery) (Experimental): Patients receive paclitaxel IV and carboplatin IV on day 1 of each cycle. Cycles repeat every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity. 6-10 weeks after cycle 1 day 1 patients undergo standard of care salvage surgery. Starting within 8 weeks of surgery, patients with high risk features also undergo radiation therapy daily for 5 treatments per week for 6 weeks and receive cisplatin IV once per week for 6 weeks during radiation treatment, in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, PET scan and optionally undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Paclitaxel; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Procedure: Salvage Surgery
- Arm 3 (Chemo-immunotherapy, salvage surgery) (Experimental): Patients receive paclitaxel IV, carboplatin IV and cemiplimab IV, over 30 minutes, on day 1 of each cycle. Cycles repeat every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity. 6-10 weeks after cycle 1 day 1 patients undergo standard of care salvage surgery. Starting within 8 weeks of surgery, patients with high risk features also undergo radiation therapy daily for 5 treatments per week for 6 weeks and receive cisplatin IV once per week for 6 weeks during radiation treatment, in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, PET scan and optionally undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Biological: Cemiplimab; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Paclitaxel; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Procedure: Salvage Surgery

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm 2 (Chemotherapy, salvage surgery); Arm 3 (Chemo-immunotherapy, salvage surgery)
Biological: Cemiplimab — Given IV
  Other Names: Cemiplimab RWLC; Cemiplimab-rwlc; Libtayo; REGN 2810; REGN-2810; REGN2810
  Arms: Arm 3 (Chemo-immunotherapy, salvage surgery)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm 2 (Chemotherapy, salvage surgery); Arm 3 (Chemo-immunotherapy, salvage surgery)
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Salvage Surgery — Undergo standard of care salvage surgery
  Other Names: Rescue Surgery; Salvage Resection; Salvage Surgical Resection; Surgical Salvage

SUMMARY:
This phase II trial tests the addition of chemotherapy, with carboplatin and paclitaxel, or chemo-immunotherapy, with carboplatin, paclitaxel and cemiplimab to standard salvage surgery followed by post operative radiation therapy and cisplatin for high risk patients, for the treatment of patients with PD-L1 positive head and neck squamous cell carcinoma that has come back and spread to nearby tissue or lymph nodes after a period of improvement (locally recurrent) or is persistent. Carboplatin is in a class of medications known as platinum-containing compounds. It works in a way similar to the anticancer drug cisplatin, but may be better tolerated than cisplatin. Carboplatin works by killing, stopping or slowing the growth of cancer cells. Paclitaxel is in a class of medications called antimicrotubule agents. It stops cancer cells from growing and dividing and may kill them. Immunotherapy with monoclonal antibodies, such as cemiplimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Salvage surgery is surgery that takes place to remove tumor tissue after a failure of other treatment. High risk patients also receive radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. Cisplatin is in a class of medications known as platinum-containing compounds. It works by killing, stopping or slowing the growth of cancer cells. Adding chemotherapy or chemo-immunotherapy to standard salvage surgery may kill more tumor cells than salvage surgery alone in patients with PD-L1 positive locally recurrent or persistent head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess and compare investigator-assessed event-free survival (EFS) of patients treated with chemotherapy (carboplatin + paclitaxel) or chemo-immunotherapy (carboplatin + paclitaxel + cemiplimab [REGN2810]) prior to salvage surgery (SS) versus patients undergoing standard of care SS.

SECONDARY OBJECTIVES:

I. To assess and compare disease-free survival (DFS). II. To assess and compare overall survival (OS). III. To assess and compare distant metastasis (DM). IV. To assess and compare acute and late toxicity (Common Terminology Criteria for Adverse Events [CTCAE] version [v] 5.0), and surgical complications.

V. To assess radiographic response (Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) to neoadjuvant therapy in the experimental arms.

VI. To assess pathologic response in the experimental arms.

EXPLORATORY OBJECTIVES:

I. To assess and compare clinical outcomes (EFS, DFS, OS, DM, and response) within the PD-L1 subgroups (combined positive score < 20 versus ≥ 20).

II. To determine the impact of surgical quality benchmarks (margin assessment, cervical lymph node harvest collected per central surgery review) and oncologic outcomes.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM 1: Patients undergo standard of care salvage surgery. Starting within 8 weeks of surgery, patients with high risk features also undergo radiation therapy daily for 5 treatments per week for 6 weeks and receive cisplatin intravenously (IV) once per week for 6 weeks during radiation treatment, in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) scan, positron emission tomography (PET) scan and optionally undergo blood sample collection throughout the study.

ARM 2: Patients receive paclitaxel IV and carboplatin IV on day 1 of each cycle. Cycles repeat every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity. 6-10 weeks after cycle 1 day 1 patients undergo standard of care salvage surgery. Starting within 8 weeks of surgery, patients with high risk features also undergo radiation therapy daily for 5 treatments per week for 6 weeks and receive cisplatin IV once per week for 6 weeks during radiation treatment, in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, PET scan and optionally undergo blood sample collection throughout the study.

ARM 3: Patients receive paclitaxel IV, carboplatin IV and cemiplimab IV, over 30 minutes, on day 1 of each cycle. Cycles repeat every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity. 6-10 weeks after cycle 1 day 1 patients undergo standard of care salvage surgery. Starting within 8 weeks of surgery, patients with high risk features also undergo radiation therapy daily for 5 treatments per week for 6 weeks and receive cisplatin IV once per week for 6 weeks during radiation treatment, in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, PET scan and optionally undergo blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 12 weeks or at the end of post operative radiation, then every 3 months for 2 years, every 6 months for years 3 and 4 and annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of locally recurrent or persistent squamous cell carcinoma of head and neck (SCCHN) arising within the oral cavity, oropharynx, larynx, or hypopharynx
* PD-L1 combined positive score (CPS) ≥ 1 using a Clinical Laboratory Improvement Amendments (CLIA) certified laboratory
* Verify insurance (or other payment) coverage for neoadjuvant chemotherapy
* Measurable disease as defined by RECIST 1.1
* Patients must have locally recurrent or persistent SCCHN arising within the oral cavity, oropharynx, larynx, or hypopharynx (American Joint Committee on Cancer [AJCC] Cancer Staging Manual, 8th Edition) AND are deemed candidates for salvage surgery:

  * P16 positive oropharynx patients with T2, T3, T4, N0, N1, N2 and all other patients with T2, T3, T4a, N0, N1, N2a, N2b, N2c, N3a are eligible.
  * Patients must be deemed surgically resectable without gross residual disease.
  * For patients with oral cavity SCCHN, only those with recurrent or persistent disease after prior surgery are eligible.
  * Patients who are candidates for salvage laryngectomy to treat recurrent laryngeal cancer and who are having salvage surgery for curative intent are eligible.
  * Patients with resectable lymph node-only recurrence are eligible.
  * No major vascular involvement (> 180° involvement of the common carotid or internal carotid artery), jugular foramen involvement, or prevertebral, paraspinous muscle involvement precluding a curative resection
* No evidence of distant metastatic disease
* The following minimum diagnostic workup is required:

  * General history and physical examination.
  * Diagnostic-quality neck CT and PET/CT of neck (PET with attenuation-correction CT of neck, chest, and abdomen)
* Age ≥ 18
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Negative urine or serum pregnancy test (in persons of childbearing potential) within 30 days prior to registration. Childbearing potential is defined as any person who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal
* Absolute neutrophil count (ANC) ≥ 1,500 cells/mm^3
* Platelets ≥ 100,000 cells/mm^3
* Hemoglobin ≥ 8.0 g/dL (Note: The use of transfusion or other intervention to achieve hemoglobin [Hgb] ≥ 8.0 g/dL is acceptable)
* Adequate renal function defined as creatinine clearance (CrCL) > 50 mL/min by the Cockcroft-Gault formula
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (Not applicable to patients with known Gilbert's syndrome)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x institutional ULN
* Only patients who received prior radiation therapy in the definitive or post-operative setting (limited to one course) are eligible.

  * Prior radiation therapy must have been completed at least 6 months prior to registration with the majority of the index persistent/recurrent cancer volume (> 50%) irradiated to ≥ 40 Gy at the time
* Prior systemic therapy including immunotherapy with anti-PD1 or anti-PDL1 within the definitive setting (neo-adjuvant, or adjuvant) is permitted and must have been completed at least 4 months prior to registration
* Prior systemic therapy including immunotherapy for treatment of recurrent or metastatic SCCHN is not permitted
* No investigational anti-cancer agents received within 4 weeks prior to registration
* No New York Heart Association Functional Classification III or IV (Note: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification)
* No active infection requiring IV antibiotics, IV antiviral, or IV antifungal treatments
* No peripheral neuropathy grade 3 or 4
* No history of allergic reaction to the study agent, compounds of similar chemical or biologic composition to the study agent, and immune checkpoint inhibitors (or any of its excipients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-10-09 (Estimated); Primary Completion 2033-02-01 (Estimated); Study Completion 2033-02-01 (Estimated)

PRIMARY OUTCOMES:
Event free survival (EFS) | From randomization to disease progression or treatment-related toxicities that precludes surgery, disease progression in the absence of surgery, disease recurrence after surgery, or death due to any cause, up to 7 years
  Will be summarized by treatment arm using standard Kaplan-Meier methods, reporting the estimated 2-year EFS rate with corresponding 95% confidence intervals.

SECONDARY OUTCOMES:
Disease free survival (DFS) | From randomization until disease recurrence, death due to any cause, up to 7 years
  Will be summarized by treatment arm using standard Kaplan-Meier methods, where estimates of the 2-year DFS will be obtained with 95% confidence intervals. Comparisons between the experimental arms and the control arm will be made using the stratified log-rank test.
Overall survival (OS) | From randomization until death due to any cause, up to 7 years
  Will be summarized by treatment arm using standard Kaplan-Meier methods, where estimates of the 2-year OS will be obtained with 95% confidence intervals. Comparisons between the experimental arms and the control arm will be made using the stratified log-rank test.
Time to distant metastasis | From randomization until detection of distant metastases or death, up to 7 years
  The cumulative incidence method will be used to estimate the incidence of distant metastases; where estimates of the 2-year distant metastasis rates will be obtained with 95% confidence intervals. Comparisons between the experimental arms and the control arm will be made using the stratified Gray's test.
Surgical complications | Up to 7 years
  Will be assessed using the Comprehensive Complication Index. Surgical complications will be summarized by treatment arm using frequencies and relative frequencies; where the overall complication rate will be estimated by treatment arm using 95% confidence intervals obtained by the Clopper-Pearson method. Comparisons between the experimental arms and the control arm will be made using the Cochran-Mantel-Haenszel test.
Incidence of acute adverse events | Up to 30 days from the last treatment
  Assessed by Common Terminology Critiera for Adverse Events (CTCAE) version (v) 5.0. The overall (highest grade) acute toxicities will be summarized by treatment arm using frequencies and relative frequencies.
Incidence of late adverse events | From day 31 to 180 days from the last treatment
  Assessed by CTCAE v 5.0. The overall (highest grade) late toxicities will be summarized by treatment arm using frequencies and relative frequencies.
Radiographic response (Arm 2 and 3) | Up to 7 years
  Response will be assessed using Response Evaluation Criteria in Solid Tumors 1.1. Best response will be summarized by treatment arm using frequencies and relative frequencies; where the complete (CR) and objective response rates (CR + partial response) will be estimated using 95% confidence intervals obtained by the Clopper-Pearson method.
Major pathological response (mPR) (Arm 2 and 3) | Up to 7 years
  mPR will be summarized by treatment arm using frequencies and relative frequencies; where the mPR rates will be estimated using 95% confidence intervals obtained by the Clopper-Pearson method.

CONTACTS AND LOCATIONS:
Overall Officials: Nabil F Saba, Principal Investigator — NRG Oncology
Locations (4):
- United States (4):
  - Sutter Medical Center Sacramento, Sacramento, California
  - Methodist Jennie Edmundson Hospital, Council Bluffs, Iowa
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm